CLINICAL TRIAL: NCT01634438
Title: Low Versus High Dose Unfractionated Heparin in Patients Undergoing Angiography Via the Radial Artery
Brief Title: Heparin Dose for Radial Angiography
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Robert Welsh, Principal Investigator, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001925
Record Dates: First submitted 2012-06-28; First posted 2012-07-06 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Angiograph
Keywords: coronary angiography
MeSH Terms: interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low dose heparin (Experimental): 30 units per kilogram of unfractionated heparin
  Interventions: Drug: unfractionated heparin
- High dose heparin (Active Comparator): 70 units per kilogram of unfractionated heparin (UFH) intravenously
  Interventions: Drug: unfractionated heparin

INTERVENTIONS:
Drug: unfractionated heparin — unfractionated heparin

SUMMARY:
At present, coronary angiogram is usually performed either through an artery in your groin or wrist. An important limitation of the wrist approach is an increase rate of blockage of the wrist artery. It is possible that the dose of blood thinner (i.e. heparin) may decrease the risk of blockage. Early studies seem to suggest that higher dose is required to reduce the risk of this important complication. However, to date there has not been a definitive study to determine the most appropriate heparin dose for the prevention of this complication. The main goal of this study is to determine the appropriate heparin dose to prevent wrist artery blockage and to determine risk factors for developing such a complication.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age who were referred for either urgent or elective cardiac catheterization were eligible for the study if a normal Allen's test was demonstrated

Exclusion Criteria:

* myocardial infarction with shock,
* ST-elevation myocardial infarction,
* patients undergoing planned percutaneous coronary intervention, and
* patients in whom transradial approach is contraindicated such as hemodialysis patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
radial artery occlusion | one month
  The primary endpoint was radial artery occlusion defined as absence palpable radial artery with no flow as assessed by Doppler study

CONTACTS AND LOCATIONS:
Locations (1):
- Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada